CLINICAL TRIAL: NCT03885739
Title: Continuous Pericapsular Nerve Group Block in Hip Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adriana Margarita Cadavid (Other)
Responsible Party: Sponsor-Investigator, Adriana Margarita Cadavid, Anesthesiologist. Specialist in Pain Medicine. Director and Clinical Professor of the Subspecialty in Pain Medicine, University of Antioquia, Universidad de Antioquia
Organization: Universidad de Antioquia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UdeA1004
Record Dates: First submitted 2019-02-27; First posted 2019-03-22 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: interventional study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with hip fracture (Other): 15 consecutive HF patients who were admitted to a single level 3 center and who report severe pain despite a standardized analgesia protocol. Patients were assessed by the Pain Service as part of a multidisciplinary care pathway and a Continuous Pericapsular Nerve Group blocks was offered as a component of a multimodal analgesic regimen.
  Interventions: Other: Continuous Pericapsular Nerve Group block

INTERVENTIONS:
Other: Continuous Pericapsular Nerve Group block — Continuous Pericapsular Nerve Group block to standardize the approach. Injections were performed using a curvilinear low-frequency ultrasound probe (3.5- to 5-MHz). The lateral border of iliopsoas tendon in an oblique axial plane at level of iliopectineal eminence provides target for needle placement. Toggling the transducer was necessary to optimize visualization of the iliopsoas tendon secondary to anisotropy. Injections were performed using an 18-gauge Tuohy needle under sterile conditions. Then, 10 mL 0.25% bupivacaine was administered and a 20-G polyamide catheter (connect to a filter) was advanced into the space. The end point of the catheter placement was the direct visualization of microbubbles in a peritendinous distribution using a bolus of agitated saline applied through threaded catheter connected to not purged filter. After catheter placement patients received a 0.1% bupivacaine continuous infusion at a constant rate.

SUMMARY:
Background- Despite clinical guidelines favoring surgical repair of hip fracture (HF) within 48 hours of injury, patients may wait considerable periods of time for their turn in the operating room. In this context, continuous nerve blocks are an attractive alternative for pain management. However, the ideal block technique is not yet defined. Recently a new ultrasound-guided approach for selective blockade of the articular branches to the hip, the PENG (Pericapsular Nerve Group) block, has been proposed with potentials advantages for perioperative hip fracture analgesia.

Objective- To describe the analgesic efficacy and feasibility of continuous Pericapsular Nerve Group block (CPENGB) in patients with HF.

Design-Interventional study. Setting-Academic Level 3 center. Methods- Two experienced anesthesiologist completed 15 sonographically guided Pericapsular Nerve Group (PENG) injections and catheter insertion in patients with severe pain awaiting HF surgery. Each injection consisted of 20 mL of local anesthetics followed by a 0.1% bupivacaine continuous infusion at a constant rate of 8 ml per hour. Pain at rest and on 15° leg lift of the fractured leg were assessed before procedure, 10 and 30 minutes after block performance, and each 24 hours until surgery. A reduction of severe or moderate dynamic pain to mild pain or no pain, and a pain relief of 2 (moderate) were clinically significant findings. To determine feasibility time and number of attempts to perform the procedure were measured.

DETAILED DESCRIPTION:
Methods: 15 sonography-guided PENG injections and catheter placement were performed in consecutive HF patients who were admitted to a single level 3 center and who report severe pain despite a standardized analgesia protocol. Patients were assessed by the Pain Service as part of a multidisciplinary care pathway and CPENGB was offered as a component of a multimodal analgesic regimen. All patients, or their legal representatives, provided written informed consent for procedure. Demographic and clinical characteristics were reviewed. To determine feasibility, time to perform the procedure was recorded, number of attempts and complications. To assess pain control, patient reported pain scores were used and the amount of morphine intravenous equivalent consumption (MIVEC) before and after block. Patients were asked to rate the severity of their pain on a 4-point numeric rating scale (Verbal Rating Scale with four response categories, VRS-4): 1) no pain, 2) mild pain, 3) moderate pain, and 4) severe pain or ''worst pain imaginable''. Pain at rest and on movement (pain on 15° leg lift of the fractured leg) were evaluated at baseline and at different times after procedure (10 minutes, 30 minutes, 24 hours and 48 hours after procedure) while the catheter was in situ. Pain relief [PR, 0 (none), 1 (slight), 2 (moderate), 3 (lots), 4 (complete)] was recorded at 30 minutes after procedure. A reduction of severe dynamic pain to mild pain or no pain, according to verbal report of patients, and a pain relief of 2 (moderate) were clinically significant findings. Type of fracture (extra or intracapsular), periprocedural complications, the presence of analgesic-related adverse effects and bromage score (30 minutes after catheter placement and each 24 hours during routine medical round) were also recorded. Complications were assessed until first orthopedic review (at 3-6 week postoperative). Procedure: All procedures were performed by two anesthesiology co-investigators who had more that 5 years of experience performing regional techniques in clinical practice and who underwent one prior training PENG blocks to standardize the approach. Injections were performed using a curvilinear low-frequency ultrasound probe (3.5- to 5-MHz). The lateral border of iliopsoas tendon in an oblique axial plane at level of iliopectineal eminence provides target for needle placement. Toggling the transducer was necessary to optimize visualization of the iliopsoas tendon secondary to anisotropy. Injections were performed using an 18-gauge Tuohy needle under sterile conditions. Following negative aspiration, a test injection was performed using 10 ml 1% lidocaine in 3-mL increments while observing in real time for ensure adequate peritendinous fluid spread of local anesthesia. Then, 10 mL 0.25% bupivacaine was administered and a 20-G polyamide catheter (connect to a filter) was advanced into the space. The end point of the catheter placement was the direct visualization of microbubbles in a peritendinous distribution using a bolus of agitated saline applied through threaded catheter connected to not purged filter. After catheter placement patients received a 0.1% bupivacaine continuous infusion at a constant rate of 8 ml per hour. If needed per anesthesiologist discretion, rescue bolus was administrated and continuous infusion rate was increased until adequate analgesia was noted. In addition, patients received a standardized analgesia protocol (preoperatively and later in the ward) consisting of 1 g paracetamol orally 2-3 times a day and opioid rescue analgesia as needed if pain moderate or severe was reported (0.05-0.1 mg/kg of intravenous morphine, or hydromorphone or tramadol equivalent, 4-6 times a day). Patients in who there were other possible causes of pain (per example: multiples traumatic lesions) received an opioid regimen by schedule plus rescue doses or intravenous patient-controlled analgesia under standardized protocols.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Acute hip fractures
* Severe pain
* Patients, or their legal representatives, provided written informed consent for procedure.

Exclusion Criteria:

* Women in pregnancy
* Trauma score greater than or equal to 16
* Incomplete data

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Verbal Rating Scale with four response categories, VRS-4 | Before procedure
  Patients were asked to rate the severity of their pain on a 4-point numeric rating scale VRS-4: 1) no pain, 2) mild pain, 3) moderate pain, and 4) severe pain or ''worst pain imaginable''. Pain at rest and on movement (pain on 15° leg lift of the fractured leg)
Verbal Rating Scale with four response categories, VRS-4 | 10 minutes after procedure
  Patients were asked to rate the severity of their pain on a 4-point numeric rating scale VRS-4: 1) no pain, 2) mild pain, 3) moderate pain, and 4) severe pain or ''worst pain imaginable''. Pain at rest and on movement (pain on 15° leg lift of the fractured leg)
Verbal Rating Scale with four response categories, VRS-4 | 30 minutes after procedure
  Patients were asked to rate the severity of their pain on a 4-point numeric rating scale VRS-4: 1) no pain, 2) mild pain, 3) moderate pain, and 4) severe pain or ''worst pain imaginable''. Pain at rest and on movement (pain on 15° leg lift of the fractured leg)
Verbal Rating Scale with four response categories, VRS-4 | 24 hours after procedure
  Patients were asked to rate the severity of their pain on a 4-point numeric rating scale VRS-4: 1) no pain, 2) mild pain, 3) moderate pain, and 4) severe pain or ''worst pain imaginable''. Pain at rest and on movement (pain on 15° leg lift of the fractured leg)
Verbal Rating Scale with four response categories, VRS-4 | 48 hours after procedure
  Patients were asked to rate the severity of their pain on a 4-point numeric rating scale VRS-4: 1) no pain, 2) mild pain, 3) moderate pain, and 4) severe pain or ''worst pain imaginable''. Pain at rest and on movement (pain on 15° leg lift of the fractured leg)

CONTACTS AND LOCATIONS:
Locations (1):
- hospital universitario San Vicente Fundacion, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Undecided